CLINICAL TRIAL: NCT01376973
Title: Efficiency of Two Occlusal Splints on TMD Treatment: Randomised Clinical Trial
Brief Title: Efficiency of Two Occlusal Splints on TMD Treatment of Police Officers
Status: Completed | Type: Observational
Sponsor: University of Campinas, Brazil (Other)
Collaborators: Coordenação de Aperfeiçoamento de Pessoal de Nível Superior. (Other Government)
Responsible Party: Paulo H. F. Caria, Unicamp
Other Study IDs: 189/03
Record Dates: First submitted 2011-06-16; First posted 2011-06-20 (Estimated); Last update posted 2011-06-20 (Estimated); Status verified 2011-06

CONDITIONS: Stress, Psychological; Temporomandibular Disorder
Keywords: stress, temporomandibular disorders.
MeSH Terms: conditions — Stress, Psychological; Temporomandibular Joint Disorders

STUDY DESIGN:
Observational Model: Case-Control | Time Perspective: Prospective
Oversight: Data Monitoring Committee: Yes

GROUPS / COHORTS (2):
- group A: Not received any oral device (Control)
- Group B and Group C: Group B - Used Michigan Occlusal Splint (MOS); Group C - Used Planas Oral Appliance (POA).

SUMMARY:
Stress is an important cause factor of temporomandibular disorder (TMD) and Police Officers are exposed to stress. Aim of the study was to evaluate clinical and electromyographically the effect of two different occlusal splints on police officers with TMD

DETAILED DESCRIPTION:
After the approval by the Human Research Ethics Committee of the Piracicaba Dental School by the register number 189/03, 905 police officers of the São Paulo State - Brazil filled up the Axis II of Research Diagnostic Criteria for Temporomandibular Disorders (RDC/TMD) and 256 volunteers were selected with TMD symptoms. Afterward the volunteers were submitted to the Axis I of RDC (clinical examination) and were excluded who presented systemic diseases like fibromyalgia, arthritis, arthrosis or osteoporosis, historical of TMJ (temporomandibular joint) surgery or TMD treatment, dental prosthesis, loss of more than two posterior teeth (except third molars and teeth extracted for orthodontic reasons), incomplete dentition with spaces in the arch (except third molars),volunteers with orthodontic and/or orthopedic appliances, with mandible and/or maxilla fractures, vertebrae or medullar canal stenosis, taking anti-inflammatory, analgesic and/or muscle-relaxing drugs, in otologic treatment or without compromise with the investigation. Who presented myogenic or mixed TMD, TMJ pain for at least three months and joint tenderness on palpation on at least one side was invited to remain in the study.

According to the exclusion and inclusion criteria above presented were selected 30 volunteers (15 women and 15 men), average age of 29 years, with diagnosis indicative of myogenic or mixed TMD.

The volunteers were randomized divided into three different groups with 10 persons per group using a stratification method performed by computerized table that placed the subjects into different groups according to the occlusal splints. Group A: Not received any oral device (Control); Group B: Used Michigan Occlusal Splint (MOS);Group C: Used Planas Oral Appliance (POA).

Each one of the 30 volunteers filled out the Visual Analog of Pain Scale (VAPS) to evaluate the muscle pain sensibility and were clinically examined according to the Axis I of RDC, always by the same examiner, in the morning, before and four weeks after the beginning of the experiment.

OCCLUSAL SPLINTS Twenty volunteers used two different occlusal splints during four weeks only while sleeping.

Volunteers were oriented to not communicate each other during treatment to keep unknown the differences between occlusal splints and about the control group.

Instrumentation Electromyographic records were performed on temporal, masseter and suprahyoid muscles before and four weeks after used the occlusal splints. Volunteers remained seated, Frankfurt's plane parallel to the floor, looking toward the front, feet on the floor, legs at 90º angle and hands resting on thighs. Occlusal splints were removed during EMG records.

All EMG records were obtained by Lynx Data Acquisition System (MCS1000-V2) with 16 channels, 12 bits resolution of dynamic range, Butterworth filter, 500 Hz pass band, high pass filter of 20 Hz and gain of 2000 times. The Software Aqdados, version 5 (Lynx) was used, with a sampling frequency of 1000 Hz and simple differential active surface electrodes with entrance impedance of 10 ohms CMRR (Common Mode Rejection Reason) of 80 dB, impedance of 1012 ohms and gain of 20 times. A reference electrode was positioned on the sternum bone of the volunteers.

Surface electrodes were placed bilaterally on the masseter, temporal and suprahyoid muscles, according to previous muscles palpation and muscle function test. In all cases electrodes were fixed on the previously cleaned skin by alcohol and attached by double-side adhesive tape (Castroflorio et al., 2004) in the centre of the muscular belly, parallel to the muscle fibers with the silver bars perpendicular to their direction to maximize signal capture and minimize noise interference.

In three different moments the EMG records were performed. First: 5 seconds of muscle resting. Second: maximal voluntary contraction (MVC), biting bilaterally two pieces of elastic cord (no.201) of 2.5-cm length. Third: MVC for the suprahyoid muscle at maximal mouth opening (MMO). Signals were normalized by the mean of the RMS (Root Mean Square) of three MVC measurements. Each EMG exam was performed after 3 minutes of resting for physiological recovery avoiding muscle fatigue.

ELIGIBILITY:
Inclusion Criteria:

* Axis II of Research Diagnostic Criteria for Temporomandibular Disorders (RDC/TMD) with TMD symptoms.

Exclusion Criteria:

* systemic diseases like fibromyalgia, arthritis, arthrosis or osteoporosis, historical of TMJ (temporomandibular joint) surgery or TMD treatment, dental prosthesis, loss of more than two posterior teeth (except third molars and teeth extracted for orthodontic reasons), incomplete dentition with spaces in the arch (except third molars),volunteers with orthodontic and/or orthopedic appliances, with mandible and/or maxilla fractures, vertebrae or medullar canal stenosis, taking anti-inflammatory, analgesic and/or muscle-relaxing drugs, in otologic treatment or without compromise with the investigation. Who presented myogenic or mixed TMD, TMJ pain for at least three months and joint tenderness on palpation on at least one side was invited to remain in the study.

Ages: 28 Years to 30 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Study Population: police officers of the São Paulo State - Brazil filled up the Axis II of Research Diagnostic Criteria for Temporomandibular Disorders (RDC/TMD) with TMD symptoms.
Sampling Method: Probability Sample
Enrollment: 30 (Actual)
Dates: Start 2008-03; Primary Completion 2008-05 (Actual); Study Completion 2008-11 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: P F Caria, PhD, Study Chair — University of Campinas - UNICAMP
Locations (1):
- University of Campinas - UNICAMP, Campinas, São Paulo, Brazil